CLINICAL TRIAL: NCT02860936
Title: Phase II Study on Lenvatinib in Recurrent and/or Metastatic Adenoid Cystic Carcinomas of the Salivary Glands of the Upper Aerodigestive Tract
Brief Title: Lenvatinib in Recurrent and/or Metastatic Adenoid Cystic Carcinomas of the Salivary Glands: ACC-LEN14
Acronym: ACC-LEN14
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 38/15
Record Dates: First submitted 2016-08-02; First posted 2016-08-10 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Adenoid Cystic Carcinomas of the Salivary Glands
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenvatinib (Experimental): 24 mg of lenvatinib will be administered daily to patients until progression of disease or intolerable toxicity or other criteria for discontinuation is met.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be self orally administered at 24 mg daily, on a continuous basis in 4 week cycles until tumour progression, unacceptable toxicity or other criteria for discontinuation is met. Study drug should be taken at approximately the same time each morning.
  Other Names: Lenvima

SUMMARY:
ACC is rare and represent approximately 25% of salivary gland carcinomas. The standard treatment is surgical excision followed by radiotherapy in selected cases. The disease is characterized by a progressive course with local and distant recurrences. First-line treatment is palliative chemotherapy that had modest results. Expression of the epidermal growth factor receptor in ACC of salivary origin has been reported. Several papers report that a high percentage of ACCs carries a chromosome translocation that results in the overexpression of the oncogene MYB, which is involved in cell proliferation, apoptosis, differentiation and in upregulation of several growth and angiogenetic factors contributing to the autocrine activation of the FGFR and VEGFR-mediated angiogenesis. Recently two whole genome sequencing of several ACC tumor/normal pairs have found mutations in genes involved in the FGF/IGF/PI3K pathway corroborating the hypothesis that this subset might benefit from inhibitors of this pathway. Based on these premises several antiangiogenic drugs and FGFR inhibitors are currently under investigation and a response rate of 11% was observed in ACC. Lenvatinib is an oral multiple RTK inhibitor targeting VEGFR-1-3, FGFR-1-4, RET, c-KIT, and PDGFR. On February 13, 2015 the drug has been approved by FDA for the treatment of patients with locally recurrent or metastatic, radioactive iodine-refractory differentiated thyroid cancer. Based on preclinical and clinical data, the investigators believe that targeting angiogenesis, FGFR pathway and tumor microenvironment might represent a rational basis to test Lenvatinib in patients with relapsed and/or metastatic ACC.

DETAILED DESCRIPTION:
Carcinomas of the salivary glands (SGCs) are rare, (less than 1% of all cancers of the head and neck and include more than 20 malignant histotypes. They can occur both in major and minor salivary glands, are locally aggressive, demonstrating invasiveness that leads to involvement of the facial nerve, skin, bone and surrounding soft tissue. The standard treatment is surgical excision, followed by radiotherapy in selected cases such as high-grade histotypes, advanced disease and neck nodes diffusion. Loco-regional recurrence occurs in 16% to 85%, it can be managed in very selected cases with further surgery and/or radiotherapy, although the prognosis of these patients remains poor. Adenoid cystic cancer (ACC) is the most common SGC histotype observed in metastatic subjects (60%) and distant metastases are the principal cause of failure, being diagnosed in 25-55% of the patients. First-line treatment is palliative chemotherapy that is typically not associated with any benefit neither in response rate nor in outcome. In preclinical models, VEGF seems to contribute to tumor aggressiveness as well as to distant metastasization, in particular in ACC. Moreover, about 80% of ACC are characterized by MYB-NFIB fusion gene. Deregulation of MYB involves several genes including those associated with apoptosis, cell cycle control and angiogenesis. Clinical evidences support the use of antiangiogenic compounds in ACC. Sorafenib a multi-tyrosine kinase inhibitor (TKI) (VEGFR1-3; PDGFR, RET, cKIT FLT3) and axitinib a potent TKI anti VEGFR1-3 have been tested in advanced ACC, obtaining a 1% of response rate, suggesting some activity agents of this class of drug.

Recently two whole genome sequencing of ACC tumor/normal pairs have found mutations in genes involved in the FGF/IGF/PI3K pathway (up to 30% of the cases) corroborating the hypothesis that this subset might benefit from agents targeting this pathway. Dovitinib, a small molecule that inhibits FGFR, is currently under investigation. Preliminary results indicate that the drug produces objective partial responses and prolonged tumor stabilization in patients with progressive ACCs. Lenvatinib has a stronger antiangiogenic effect compared to sorafenib and axitinib and has also a higher potency with regard to inhibition of FGFR-1, offering a potential opportunity to block one of the well known mechanisms of resistance to VEGF/VEGFR inhibitors. Lenvatinib also has a direct oncogenic effect of controlling tumor cell proliferation by inhibiting RET, c-KIT, and PDGFR beta, as well as an effect on the tumor microenvironment by blocking FGFR and PDGFR beta.

Lenvatinib has been investigated in thyroid cancer and hepatocellular carcinoma (phase III trials) and in other malignancies, showing high rates of activity.

Based on preclinical and clinical data, the investigators believe that targeting angiogenesis, FGFR pathway and tumor microenvironment might represent a rational basis to test lenvatinib in patients with relapsed and/or metastatic ACC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven relapsed and/or metastatic adenoid cystic carcinoma for which potentially curative options such as surgery or radiotherapy are not indicated.
2. Archival tissue samples or unstained 20 slides from primary tumor or metastasis for translational biological research.
3. Subjects with at least one uni-dimensional measurable lesion by CT-scan or MRI according to RECIST criteria 1.1 (target lesion). A previously treated lesion by radiotherapy or loco-regional therapies such as radiofrequency (RF) can be chosen as target lesion only if progression in the respective lesion has been demonstrated during or following radiotherapy.
4. Clinical or radiological progression of disease within 6 months at study entry. Progression of disease by RECIST is not required.
5. Age ≥ 18 years
6. ECOG Performance Status < 2
7. Life expectancy of > 3 months
8. Adequately controlled blood pressure with or without antihypertensive medications, defined as BP < 150/90 mmHg at screening and no change in antihypertensive medications within 1 week prior to Cycle 1 Day 1
9. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

   * Hemoglobin >9.0 g/dl
   * Neutrophil count (ANC) >1,000/mm3
   * Platelet count 75,000/μl
   * Total bilirubin <1.5 times the upper limit of normal
   * ALT and AST <2.5 x upper limit of normal (<5 x upper limit of normal for patients with liver metastases)
   * Serum creatinine <1.5 x upper limit of normal
   * Alkaline phosphatase <4 x ULN
   * PT-INR/PTT <1.5 x upper limit of normal (Patients who are being therapeutically anticoagulated with an agent such as heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists)
10. Previous systemic therapy for metastatic disease is allowed for a maximum of 1 previous line of chemotherapy and/or 1 previous line of TKI
11. Signed written informed consent

Exclusion Criteria:

1. Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry
2. Subjects having > 1+ proteinuria on urine dipstick testing will undergo 24h urine collection for quantitative assessment of proteinuria. Subjects with urine protein ≥ 1 g/24h will be ineligible
3. History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
4. Gastrointestinal abnormalities (i.e. inability to take oral medication; malabsorption syndrome)
5. Requirement for anticoagulant therapy with oral vitamin K antagonists (LMWH therapy is accepted)
6. Prolongation of QTc interval to > 480 msec
7. Known allergic reaction to any of the components of the treatment
8. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
9. Legal incapacity or limited legal capacity
10. Active clinically serious infections (> grade 2 NCI-CTC version 4.0)
11. Medical or psychological condition which, in the opinion of the investigator, would not enable the patient to complete the study or knowingly sign the Informed Consent
12. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and two weeks after the completion of trial
13. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
14. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
15. History of organ allograft.
16. Patients with evidence or history of bleeding diathesis
17. Patients undergoing renal dialysis
18. Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry.
19. Previous therapy with lenvatinib (E7080)
20. Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy will be allowed)
21. Major surgery within 2 weeks of start of study
22. Use of biologic response modifiers, such as G-CSF, within 3 week of study entry [G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator, however they may not be substituted for a required dose reduction; patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study]
23. Investigational drug therapy outside of this trial during or within 4 weeks of study entry

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-06; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate (CR+PR) | 2 years and 5 months
  Objective response rate (CR+PR) will be evaluated according to RECIST response evaluation criteria 1.1 at any subsequent re-evaluation

SECONDARY OUTCOMES:
Progression free survival | 2 years and 5 months
  PFS according to RECIST criteria 1.1
Overall survival | 2 years and 5 months
  After study drug treatment ends, patients will be contacted each 6 months to determine survival
Safety and toxicity profile of lenvatinib (according to CTCAE v 4.0) | 2 years and 5 months
  Incidence of adverse events (AEs), will be graded according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.0, laboratory values, physical examinations, vital signs.
Duration of response | 2 years and 5 months
  The duration of response will be evaluated to assess the duration of activity of lenvatinib (CR+PR+SD)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Only study results will be shared through publication on scientific indexed journals

REFERENCES:
- [Derived] Locati LD, Galbiati D, Calareso G, Alfieri S, Singer S, Cavalieri S, Bergamini C, Bossi P, Orlandi E, Resteghini C, Platini F, Granata R, Quattrone P, Mancinelli M, Mariani L, Lo Vullo S, Licitra LF. Patients with adenoid cystic carcinomas of the salivary glands treated with lenvatinib: Activity and quality of life. Cancer. 2020 Jan 1;126(9):1888-1894. doi: 10.1002/cncr.32754. Epub 2020 Feb 7. PMID 32031693